CLINICAL TRIAL: NCT06121934
Title: Efficacy and Safety of Carica Papaya in Dengue Fever: A Randomised Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Collaborators: Institute of Technology Transfer and Innovation (ITTI) (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Shohael Mahmud Arafat, Professor, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BSMMU/2023/12097
Record Dates: First submitted 2023-10-24; First posted 2023-11-08 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Dengue
Keywords: Dengue fever; severity reduction; carica papaya; CPLE; RCT
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Intervention Model Description: Two arms are being used in this study, One arm contains active drug and other contains placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The recruiter, caregiver, randomizer, and investigator all are blinded, except for the manufacturer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carica Papaya Leaf Extract (Experimental): The study patients will be followed for clinical and laboratory endpoints in the hospital until study day 5 (or daily as outpatients from discharge to day 5) and reviewed at an outpatient visit at week 2 after discharge.
  The patients will be assigned to one of the two treatment arms after randomization:
  1) Active drug: Carica papaya leaf extract (CPLE) 500mg 2 capsule t.i.d for 5 days
  The oral capsule of CPLE and placebo will be provided by the Institute of Technology Transfer and Innovation (ITTI), an institute in Bangladesh Council of Scientific and Industrial Research (BCSIR), with appropriate masking for a double-blind study. On receipt, the medications will be stored in a secure area by the manufacturer's recommendation.
  Interventions: Drug: Carica Papaya Leaf Extract
- Placebo (Placebo Comparator): The study patients will be followed for clinical and laboratory endpoints in the hospital until study day 5 (or daily as outpatients from discharge to day 5) and reviewed at an outpatient visit at week 2 after discharge.
  The patients will be assigned to standard treatment with placebo after randomization:
  Placebo: visually matched placebo 2 capsule t.i.d for 5 days
  The oral capsule of CPLE and placebo will be provided by the Institute of Technology Transfer and Innovation (ITTI), an institute in Bangladesh Council of Scientific and Industrial Research (BCSIR), with appropriate masking for a double-blind study. On receipt, the medications will be stored in a secure area by the manufacturer's recommendation.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carica Papaya Leaf Extract — Active drug: CPLE 500mg 2 capsule t.i.d for 5 dayseive CPLE or placebo once daily for 5 days.
  Arms: Carica Papaya Leaf Extract
Drug: Placebo — Placebo: visually matched placebo 2 capsule t.i.d for 5 days
  Arms: Placebo

SUMMARY:
This will be a placebo-controlled, multicenter-randomized prospective study of CPLE (Carica papaya leaf extract) tabs in dengue patients (WHO-Group A, B). The study will enroll 300 eligible dengue cases into two arms: one arm receiving CPLE 1000mg t.i.d for 5 days and the other group receiving a placebo.

The main question to ask is whether CPLE reduces severe disease progression and increases platelet counts in dengue patients.

The participant will be asked to take orally available CPLE capsules at a dose of 1000 mg (2 capsules, 500mg each) or identical placebo three times a day for 5 days

DETAILED DESCRIPTION:
Introduction:

Dengue is the most important emerging viral disease of humans that, in recent decades, has become a major international public health concern. Dengue is found in tropical and subtropical regions worldwide, predominantly in urban and semi-urban areas. Dengue infection is transmitted through Aedes agypti, a Flaviviridae virus . Dengue occurs within 5-7 days after an infected mosquito bites a healthy person. There is no specific treatment for dengue; intensive supportive care is the most important aspect of management. The thrombocytopenia which usually happens in the defervescence stage of the illness is the critical phase, and if left unattended or untreated it can lead to mortality. Till now there is no approved vaccine or drug against dengue virus, therefore there is an urgent need of development of alternative solutions for dengue. Several plants species have been reported with anti-dengue activity. Researchers have indicated that the juice of the leaves of the Carica papaya plant from the family Caricaceae helps to increase the platelet levels and have demonstrated definitive beneficial effects in these patients.Carica papaya leaf extract can be used in any form for its ability on three aspects of dengue: antiviral activities, prevention of thrombocytopenia and improvement of immunity during dengue fever. Papaya leaf extract being a strong stimulant of IL-6 and SCF might help to improve thrombocytopenic conditions of the infected patients. Papaya leaves extract, rich in papain, was shown to improve thrombocyte (platelet) count in dengue patients. The qualitative phytochemical analysis reveals that except steroids and tannins all the phytochemical including glycosides, alkaloids, saponins, flavonoids, proteins are present in leaf of papaya. Papaya leaf contains anti-oxidant vitamins and minerals which may help to increase the hemoglobin,hematocrit, Red blood cells, thrombocytes and total protein contents.

Rationale:

Since there is no antiviral or vaccine to prevent dengue infections, symptomatic and supportive care must be used as the main forms of treatment. Although their effectiveness in such circumstances is debatable, prophylactic, or therapeutic platelet transfusions occasionally treat dengue-induced thrombocytopenia with or without significant hemorrhagic symptoms. Additionally, many patients find processing platelet transfusion expensive, and this platelet separation machine is unavailable in many distant places. There are several reports of using natural treatments to treat dengue thrombocytopenia. In several nations, oral administration of the extraction of Carica papaya leaves is used as a natural antipyretic treatment for dengue fever with thrombocytopenia. This extract has been shown in several experimental investigations both preclinical and clinical to have the ability to stabilize erythrocytes and stop hemolysis. Additionally, it has been demonstrated to directly influence platelets by blocking their aggregation, particularly during dengue infections. It has been demonstrated that CPLE increases platelet counts in patients with mild to moderate thrombocytopenia safely and effectively. It has not yet been determined how effective CPLE is at reducing the severity of dengue fever and the reduction of severe thrombocytopenia brought on by dengue. In this trial, the investigators want to find out the effectiveness and safety of CPLE in treating dengue patients by reducing severe progression, increasing platelet counts, and lowering the requirement for platelet transfusions.

Research question: Is CPLE effective in treating dengue patients by reducing severe disease progression and increasing platelet counts?

Research Hypothesis:

Null hypothesis: There is no difference in efficacy between CPLE and placebo in reducing severe disease progression and increasing platelet counts in patients with dengue fever.

Alternative hypothesis: CPLE is more effective than placebo in reducing severe disease progression and increasing platelet counts in patients with dengue fever.

Objectives:

Primary Objective: To determine the efficacy of CPLE in the reduction of severe disease progression and increasing platelet count in dengue patients.

Secondary Objectives:

1. To see the efficacy of CPLE in reduction of severe disease progression in dengue patients
2. To find out the efficacy of CPLE in increasing platelet count in dengue patients
3. To observe any bleeding episodes in hospitalized dengue patients between the CPLE and placebo group
4. To explore the side effect profile of CPLE in treating dengue patients
5. To observe reduction in the number of transfusions of all blood products, including platelets
6. To find out the total length of hospital (ICU & ward) stay between the groups
7. Reduction of all causes of mortality in dengue patients

Study Outcome Measures Primary endpoint The major effectiveness endpoints will be determined by comparing the rise in platelet counts and normalization of hematocrit levels between the treatment and placebo groups during the hospital stay. The treatment and placebo groups will also compare the peak platelet count and normalization of hematocrit value. The two trial groups will also compare the disease severity progression also, frequency and kind of blood products-especially platelet transfusions-needed to treat thrombocytopenia during illness.

Secondary endpoint The secondary outcomes the investigators plan to evaluate include parameters indicative of disease progression between the two study arms.

1. The frequency of bleeding events determined by clinical evaluation twice daily will also be compared between the treatment and placebo groups. Evidence of internal organ bleeding, hypotension, small mucosal hemorrhages, sub-conjunctival hemorrhages, epistaxis, petechiae or ecchymosis, hematemesis, cerebral bleeding, and melena will be evaluated.
2. The type of bleeding manifestation between the two arms of the study will be characterized. The investigators will examine the evidence of (mucosal, GI, GU, vaginal, IC bleed, etc.) bleeding with the severity of thrombocytopenia and response to intervention by comparing both arms.
3. Safety and tolerability will also be assessed by comparing the proportion of patients who experience any AE (adverse event) and any SAEs between the treatment arms.
4. To correlate the change in platelet counts and subsequent response with or without CPLE (Caripill) to the phase of dengue (febrile/critical/ convalescent). Additionally, the investigators will compare both arms of the study to examine if the intervention in any of the three phases affected the duration/severity of thrombocytopenia.
5. Date of admission and date of discharge or death will be noted in the CRFs and will be used to determine the length of hospital stay (ICU & Ward), in dengue patients receiving CPLE (Caripill) treatment compared to the placebo group.

Materials and method:

Study design: Randomized double-blind placebo-controlled multicenter prospective trial Period of study: September 2023 to February 2024 Place of study: Department of Internal Medicine, BSMMU Study population: Any patient with dengue fever

ELIGIBILITY:
Inclusion Criteria:

* Patients who are confirmed dengue fever by NS1 dengue Ag or anti dengue Ab IgM positive

Exclusion Criteria:

* Children (<18 years)
* Currently pregnant or lactating
* Patients on steroids, any immunosuppressant
* Patients who received platelet transfusion during the same admission
* Patient with other known causes of thrombocytopenia, including leukemia, ITP
* Patients with alanine aminotransferase (ALT) levels >150 U/L
* Patient with serum creatine >1.4 mg/dl
* S. creatine kinase (CK) >1000 U/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Rise in platelet counts | Within five days
  The treatment and placebo groups will compare the peak platelet count
Return of hematocrit levels towards baseline | Within five days
  The treatment and placebo groups will compare the normalization of hematocrit value

SECONDARY OUTCOMES:
Bleeding Manifestations | Within six days
  The frequency of bleeding events determined by clinical evaluation between the treatment and placebo groups
Duration of hospital stay | Within six days
  Admission and date of discharge or death will be noted in the case record form and will be used to determine the length of hospital stay between the active and placebo groups

CONTACTS AND LOCATIONS:
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after completion of study

REFERENCES:
- [Background] Ahmad N, Fazal H, Ayaz M, Abbasi BH, Mohammad I, Fazal L. Dengue fever treatment with Carica papaya leaves extracts. Asian Pac J Trop Biomed. 2011 Aug;1(4):330-3. doi: 10.1016/S2221-1691(11)60055-5. PMID 23569787
- [Background] Subenthiran S, Choon TC, Cheong KC, Thayan R, Teck MB, Muniandy PK, Afzan A, Abdullah NR, Ismail Z. Carica papaya Leaves Juice Significantly Accelerates the Rate of Increase in Platelet Count among Patients with Dengue Fever and Dengue Haemorrhagic Fever. Evid Based Complement Alternat Med. 2013;2013:616737. doi: 10.1155/2013/616737. Epub 2013 Apr 11. PMID 23662145
- [Background] Kasture PN, Nagabhushan KH, Kumar A. A Multi-centric, Double-blind, Placebo-controlled, Randomized, Prospective Study to Evaluate the Efficacy and Safety of Carica papaya Leaf Extract, as Empirical Therapy for Thrombocytopenia associated with Dengue Fever. J Assoc Physicians India. 2016 Jun;64(6):15-20. PMID 27739262
- [Background] Sarker MMR, Khan F, Mohamed IN. Dengue Fever: Therapeutic Potential of Carica papaya L. Leaves. Front Pharmacol. 2021 Apr 26;12:610912. doi: 10.3389/fphar.2021.610912. eCollection 2021. PMID 33981215